CLINICAL TRIAL: NCT04743323
Title: A Case-CrossovEr Study deSign to Inform Tailored Interventions to Prevent Disease
Brief Title: A Case-CrossovEr Study deSign to Inform Tailored Interventions to Prevent Disease Progression in Acute Pancreatitis
Acronym: ACCESS-AP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Pittsburgh (Other); Alcohol Research Group (Other); Ohio State University (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christie Jeon, Research Scientist, Cedars-Sinai Medical Center
Other Study IDs: STUDY00000364; 7W81XWH1910888 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pancreatitis, Acute; Alcohol Drinking; Health Behavior
MeSH Terms: conditions — Pancreatitis; Alcohol Drinking; Health Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants will be recruited whilst hospitalized for an acute episode of pancreatitis. They will be interviewed about their health behaviors including alcohol consumption during the two weeks immediately preceding the onset of pancreatitis. Blood and urine bio-specimens will be collected at this time.
  Following discharge from hospital (5-26 weeks) the same participant will be interviewed again during an asymptomatic control period and blood and urine bio-specimens will be collected. This study will compare the participant's exposure immediately preceding the onset of pancreatitis to that of an asymptomatic control period from the same participant.
  Participants will be followed for 24 months via review of their medical records every 6 months to assess any recurrent disease or progression of disease.

SUMMARY:
The Purpose of this study is to investigate changes in alcohol consumption in the period leading up to the onset of pancreatitis and compare that to levels of drinking during asymptomatic periods.

DETAILED DESCRIPTION:
There is no question that long-term heavy consumption of alcohol leads to increased risk of recurrent acute and chronic pancreatitis. While many patients and providers assume that heavy episodic alcohol consumption leads to acute pancreatitis, it is yet unknown whether 'binge' drinking truly causes pancreatitis and if so, what the relevant timing and duration of hazardous alcohol consumption is. Because of the lack of clarity on the transient effects of alcohol on acute pancreatitis, patients and providers are left with an uncertain disease progression and lack of tailored alcohol reduction recommendations.

Our study aims to investigate changes in alcohol consumption in the period leading up to the onset of pancreatitis and compare that to levels of drinking during asymptomatic periods. This epidemiologic design is called the case-crossover study, in which the diseased person serves as his/her own control. This study design has advantages over typical case-control studies in that factors that do not change within the individual, such as sex, race, genetic risks, will not interfere with evaluating the causal role of heavy episodic drinking on pancreatitis.

Participants in this study will undergo detailed interview on recent and lifetime alcohol consumption and other correlated health behaviors while they are hospitalized. Blood and urine will be collected during the hospitalization. After discharge, they will be interviewed again for any changes in alcohol consumption and blood and urine will be collected during a standard of care visit. The investigators will chart the progression of their disease through quarterly check-up by phone and through the medical records.

Ultimately, the investigators aim to generate data that will empower patients and providers to develop tailored regimens for prevention of recurrent acute pancreatitis, that will have lasting beneficial effects in averting irreversible damage to the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years at the time of eligibility assessment
* Currently hospitalized with Acute Pancreatitis (AP) per Revised Atlanta Classification, which requires two of the following evidence of pancreatitis:

  1. Abdominal pain consistent with AP (acute onset of a persistent, severe, epigastric pain often radiating to the back)
  2. Serum lipase activity (or amylase activity) at least three times greater than the upper limit of normal
  3. Characteristic findings of AP on computed tomography (CT), magnetic resonance imaging (MRI) or transabdominal ultrasonography
* Alcohol Use Disorders Identification Test Consumption (AUDIT-C) alcohol consumption score of ≥3

Exclusion Criteria:

* Pancreatitis presumed to be related to: gallstones, medication, trauma, autoimmune pancreatitis, post-ERCP pancreatitis, pancreatic ductal adenocarcinoma, suspected cystic neoplasm, neuroendocrine tumors, and other uncommon tumors.
* Chronic pancreatitis with calcification(s).
* Pancreatic cancer or pancreatic metastasis from other malignancies.
* History of pancreas transplant or pancreatectomy
* Current medical or psychiatric illnesses that in the investigator's opinion would compromise their ability to tolerate study procedures or participate in longitudinal follow up.
* Currently incarcerated.
* Known current pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults that consume alcohol who are hospitalized for acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | Between 5-26 weeks
  Compare alcohol consumption prior to an attack of Acute Pancreatitis to that during an asymptomatic control period. Alcohol consumption will be measured by a 48-hour recall questionnaire, and timeline follow-back instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Christie Y Jeon, ScD, Principal Investigator — Cedars-Sinai Medical Center
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Ohio State University, Columbus, Ohio
  - University of Pittsburg, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cherpitel CJ, Ye Y, Bond J, Borges G, Macdonald S, Stockwell T, Room R, Sovinova H, Marais S, Giesbrecht N. Validity of self-reported drinking before injury compared with a physiological measure: cross-national analysis of emergency-department data from 16 countries. J Stud Alcohol Drugs. 2007 Mar;68(2):296-302. doi: 10.15288/jsad.2007.68.296. PMID 17286349
- [Background] Jeon CY, Papachristou GI, Pisegna JR, Pendergast FJ, Lin YC, Cherpitel CJ, Ye Y, Pandol SJ, Yadav D. A Case-CrossovEr study deSign to inform tailored interventions to prevent disease progression in Acute Pancreatitis (ACCESS-AP) - study design and population. Pancreatology. 2021 Oct;21(7):1231-1236. doi: 10.1016/j.pan.2021.06.007. Epub 2021 Jun 24. PMID 34229971
- [Result] Jeon CY, Adeniran E, Stewart C, Papachristou GI, Pisegna JR, Kuc AA, Buxbaum JL, Pandol SJ, Yadav D. Female patients delay seeking medical care with alcohol-associated acute pancreatitis. Pancreatology. 2023 Nov;23(7):761-766. doi: 10.1016/j.pan.2023.08.001. Epub 2023 Aug 5. PMID 37567847